CLINICAL TRIAL: NCT07379112
Title: A Prospective, Multi-centre, Single-arm Registry to Evaluate the Safety and Performance of Dafodil™ Pericardial Bioprosthesis Series in Participants Undergoing Native/Prosthetic Aortic or Mitral Valve Replacement in Real World Settings
Brief Title: Safety and Performance of Dafodil Heart Valves in Real-World Aortic and Mitral Valve Replacement
Status: Not yet recruiting | Type: Observational
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLS/EURODAF-1; MLS/EURODAF-1 (Other: Meril Life Sciences Pvt. Ltd.)
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Disease, Mitral Valve Disease, Prosthetic Heart Valve Dysfunction; Valvular Heart Disease Requiring Surgical Aortic or Mitral Valve Replacement
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgical aortic or mitral valve replacement with the Dafodil™ or Dafodil Neo™ pe: Participants undergoing surgical replacement of a native or failed prosthetic aortic or mitral valve using the Dafodil™ or Dafodil Neo™ pericardial bioprosthetic heart valve. Participants are followed prospectively to assess safety and performance outcomes in real-world clinical practice.
  Interventions: Device: Dafodil™ / Dafodil Neo™ Pericardial Bioprosthetic Heart Valve

INTERVENTIONS:
Device: Dafodil™ / Dafodil Neo™ Pericardial Bioprosthetic Heart Valve — The Dafodil™ and Dafodil Neo™ pericardial bioprosthetic heart valves are surgically implanted for replacement of a diseased or failed native or prosthetic aortic or mitral valve as part of standard clinical care. This observational registry prospectively follows participants to evaluate the safety and performance of the device in real-world clinical practice.

SUMMARY:
This study, called the EuroDafodil Registry, is being conducted to understand how safe and effective the Dafodil™ and Dafodil Neo™ Pericardial Bioprosthetic heart valves are when used in routine medical practice.

The registry includes adult patients (18 years or older) who require surgical replacement of their aortic or mitral heart valve, either because their natural valve is severely diseased or because a previously implanted valve is no longer working properly. All patients in this registry will receive a Dafodil™ heart valve as part of their standard surgical treatment. No experimental procedures are involved beyond usual clinical care.

This is a prospective, multi-centre registry being conducted at approximately 50 hospitals across Europe, with a planned enrollment of at least 500 patients. The study does not compare treatments; instead, it follows patients who receive the Dafodil™ valve to collect real-world information on outcomes.

Doctors will monitor patients during their hospital stay and through regular follow-up visits at 1 or 3 months, 1 year, 3 years, and up to 5 years after surgery. Information collected includes survival, heart valve function, complications such as blood clots or infections, heart performance on echocardiography, and quality of life.

Participation in this registry is voluntary. All patients must provide written informed consent before joining. Patient privacy will be protected: personal identifiers will not be shared, and data will be coded so individuals cannot be directly identified.

The results of this registry will help doctors and health authorities better understand the long-term safety, performance, and durability of the Dafodil™ heart valves in real-world clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥18 years of age
* Participants whose valvular disease is sufficiently advanced to warrant replacement of their natural/prosthetic aortic or mitral valve with Dafodil pericardial bioprosthesis series
* Participants who are willing to undergo all protocol specific study procedures and follow-up requirements

Exclusion Criteria:

* Participants who are not willing to provide informed consent form, or whose legal heirs object to their participation in the registry
* Participant with active endocarditis, active myocarditis or other systemic infection
* Participants undergoing double valve replacement (DVR)
* Any condition, which, in Investigator's opinion would preclude safe participation of participants in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced aortic or mitral valvular heart disease undergoing surgical replacement of a native or failed prosthetic valve with a bioprosthetic heart valve in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Mortality, Thromboembolism, Valve Thrombosis, Paravalvular Leak, and Endocarditis | 1 year
  Composite of all-cause mortality, thromboembolism, valve thrombosis, major paravalvular leak, and endocarditis following surgical aortic or mitral valve replacement with a bioprosthetic heart valve.